CLINICAL TRIAL: NCT01965899
Title: Reveal LINQ Usability Study
Brief Title: Usability Study to Assess the Reveal LINQ Insertable Cardiac Monitor System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Reveal LINQ Usability Study
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Results first posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-06

CONDITIONS: Syncope; Recurrent Symptomatic Atrial Fibrillation
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insertable Cardiac Monitor Implant (Experimental)
  Interventions: Device: Insertable Cardiac Monitor Implant

INTERVENTIONS:
Device: Insertable Cardiac Monitor Implant — The Reveal LINQ is a leadless device that is recommended to be implanted in the region of the thorax. Two electrodes on the body of the device continuously monitor the patient's subcutaneous ECG. The device stores ECG recordings from the patient-activated episodes and ECG recordings from automatically detected arrhythmias. Documentation of episode occurrence will be retained.

SUMMARY:
The purpose of the Reveal LINQ Usability Study is to assess the functionality of the Reveal LINQ insertable cardiac monitor and accompanying system in patients indicated for an insertable cardiac monitor

DETAILED DESCRIPTION:
The Reveal LINQ Usability Study is a prospective, non-blinded, non-randomized, multi-center clinical trial. Subjects will transmit device data via manual interrogation on a weekly basis during the first month and will be evaluated in the office at 1-month post-implant, in addition to an automatic nightly wireless data transmission using the MyCareLink® home monitor. All subjects will be requested to wear an external Holter for 48 hours at approximately 4 weeks post-insertion. Follow-up visits will continue at 6 and 12 months post-implant, with monthly manual interrogations. Subjects will be exited at their 12 month follow-up visit. The overall study will be conducted in 2 phases which differ primarily on inclusion criteria: Phase I subjects (initial 30 subjects) will have any indication for an ICM, Phase II subjects (all subjects following the initial 30 subjects) will be atrial fibrillation (AF) pre-ablation patients. The study will assess functionality of the Reveal LINQ device by assessing sensing performance and data transmission.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to sign and date the consent form.
* Subject is indicated for a Reveal device within the existing market approved indications
* Phase I (initial 30 subjects): Any indication for a Reveal LINQ Device
* Phase II (after the initial 30 subjects): Subject has atrial fibrillation and is indicated for and identified as an AF pre-ablation candidate*

  *Note: Atrial fibrillation must be documented in the subject's medical history.
* Subject has a life expectancy of 18 months or more.
* Subject is willing and able to set up and utilize MyCareLink® home monitor and be remotely monitored (i.e., Medtronic CareLink® Network)
* Subjects who are female of childbearing potential (last menses less than 1 year prior to enrolment) must:
* have a negative pregnancy test at enrollment.
* not be breastfeeding.
* either be surgically sterile, postmenopausal (cessation of menses for at least 1 year), or agree to use a medically accepted, highly effective method of contraception during the entire duration of the study.

Exclusion Criteria:

* Subject has an active implanted cardiac medical device (e.g., IPG, ICD, CRT, etc).
* Subject is unwilling or unable to comply with the study procedures
* Subject is legally incapacitated and unable to provide written informed consent.
* Any concomitant condition which, in the opinion of the investigator, would not allow safe participation in the study (e.g., drug addiction, alcohol abuse, emotional/psychological diagnosis)
* Patient is enrolled in another study that could confound the results of this study, without documented pre-approval from Medtronic study manager.
* Local law prohibits participation (e.g., minor status as specified by local law)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Pürerfellner, MD, Principal Investigator — Allgemein öffentliches Krankenhaus der Elisabethinen Linz; Lukas Dekker, MD, Principal Investigator — Catharina Ziekenhuis
Locations (16):
- Australia (3):
  - The Prince Charles Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria
- Austria (2):
  - Allgemein öffentliches Krankenhaus der Elisabethinen Linz, Linz
  - Allgemeines Krankenhaus der Stadt Linz, Linz
- Belgium (2):
  - UZ Leuven - Campus Gasthuisberg, Leuven
  - CHU UCL Mont-Godinne - Dinant, Yvoir
- Netherlands (5):
  - Catharina Ziekenhuis, Eindhoven
  - Academisch Ziekenhuis Maastricht, Maastricht
  - St. Antonius Ziekenhuis - Locatie Nieuwegein, Nieuwegein
  - Diakonessenhuis Locatie Utrecht, Utrecht
  - Isala Klinieken - Locatie Weezenlanden, Zwolle
- Scientific Research Institute of Circulation's Pathology Agency on High Medical Technologies, Novosibirsk, Russia
- Narodny ustav srdcovych a cievnych chorob, a.s. (NUSCH), Bratislava, Slovakia
- United Kingdom (2):
  - Eastbourne District General Hospital, Eastbourne
  - James Cook University Hospital, Middlesbrough

REFERENCES:
- [Derived] Saiz-Vivo J, Abdollahpur M, Mainardi LT, Corino VDA, De Melis M, Hatala R, Sandberg F. Heart rate characteristic based modelling of atrial fibrillatory rate using implanted cardiac monitor data. Physiol Meas. 2023 Mar 10;44(3). doi: 10.1088/1361-6579/acbc08. PMID 36787645
- [Derived] Purerfellner H, Sanders P, Pokushalov E, Di Bacco M, Bergemann T, Dekker LR; Reveal LINQ Usability Study Investigators. Miniaturized Reveal LINQ insertable cardiac monitoring system: First-in-human experience. Heart Rhythm. 2015 Jun;12(6):1113-9. doi: 10.1016/j.hrthm.2015.02.030. Epub 2015 Feb 26. PMID 25728756

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insertable Cardiac Monitor Implant
Started | 151
Completed | 145
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Insertable Cardiac Monitor Implant
Number analyzed (Participants) | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 101
Region of Enrollment [Number; unit: participants]
  Russian Federation | 7
  Netherlands | 40
  Austria | 28
  Belgium | 10
  United Kingdom | 8
  Slovakia | 25
  Australia | 33

OUTCOME MEASURES:

1. Primary Outcome: Success of Wireless Transmissions
Description: To assess the percentage of successful automatic wireless transmissions from the system within the first 30 days of implant.
Time Frame: 30 days
Population: All 151 subjects received a CareLink monitor software update. Subjects contributed 4,511 follow-up days in their first 30 days.
Measure: Number (95% Confidence Interval); unit: percentage of successful transmissions
Units Other Than Participants: Automatic Transmissions
Arm/Group | Insertable Cardiac Monitor Implant
Number analyzed (Participants) | 151
Number analyzed (Automatic Transmissions) | 4511
percentage of successful transmissions | 73.1 [68.3 to 77.4]

2. Primary Outcome: R-wave Amplitude
Description: To characterize the signal quality of the R-wave amplitude at implant and one month.
Time Frame: 30 days
Population: For each subject implanted with a Reveal LINQ device an R-wave amplitude measurement is collected at implant and 1 month follow-up.
Measure: Mean (Standard Deviation); unit: μV
Arm/Group | Insertable Cardiac Monitor Implant
Number analyzed (Participants) | 151
μV
  R-wave at implant (n=151) | 543.5 (294.8)
  R-wave at one month follow-up (n=150) | 599.4 (314.2)

3. Primary Outcome: R-wave Amplitudes Greater Than or Equal to 200 μV
Description: The proportion of R-wave amplitudes that are greater than or equal to 200 μV will be estimated at implant and one month.
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: Percentage of subjects
Arm/Group | Insertable Cardiac Monitor Implant
Number analyzed (Participants) | 151
Percentage of subjects
  Implant | 97.3
  1 Month | 96.6

4. Secondary Outcome: Accuracy of Reveal LINQ Device Detected Atrial Fibrillation
Description: To assess atrial fibrillation detection by the Reveal LINQ insertable cardiac monitor (ICM). True and false positives will be reported.
Time Frame: 4 months
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes
Arm/Group | Insertable Cardiac Monitor Implant
Number analyzed (Participants) | 151
Number analyzed (Episodes) | 5304
Episodes
  True positive | 4461
  False positive | 843

5. Secondary Outcome: Safety Endpoint
Description: To characterize the system-related and procedure-related adverse events.
Time Frame: 12 months
Measure: Number; unit: Number of events
Arm/Group | Insertable Cardiac Monitor Implant
Number analyzed (Participants) | 151
Number of events
  Procedure related | 9
  System related | 45
  Procedure related (Serious events) | 1
  System related (Serious events) | 1

6. Secondary Outcome: Accuracy of Device Detected Atrial Fibrillation Compared to Holter Monitor
Description: To compare the Reveal LINQ atrial fibrillation detection accuracy with atrial fibrillation detection from Holter monitoring. The true positive rate (sensitivity), specificity, positive predictive value and negative predictive value will be estimated using Holter recordings as the gold standard. Sensitivity measures the proportion of positives that are correctly identified as such. Specificity measures the proportion of negatives that are correctly identified as such. The positive and negative predictive values are the proportion of positive and negative detected patients that are true positive and true negative, respectively. Accuracy measures the proportion of all patients that are correctly identified as negative or positive.
Time Frame: 48 hours
Population: A Holter recording was performed in all 150 patients (one patient exited before 1 month), of which 141 were suitable for analysis after excluding recordings with technical issues, such as loss of telemetry or inability to process the data.
Measure: Number; unit: Percentage of patients
Groups:
- Insertable Cardiac Monitor Implant: The Reveal LINQ is a leadless device that is recommended to be implanted in the region of the thorax. Two electrodes on the body of the device continuously monitor the patient's subcutaneous ECG. The device stores ECG recordings from the patient-activated episodes and ECG recordings from the automatically detected arrhythmias. Documentation of episode occurrence will be retained.
Arm/Group | Insertable Cardiac Monitor Implant
Number analyzed (Participants) | 141
Percentage of patients
  Sensitivity | 97.4
  Specificity | 97.0
  Positive predictive value | 92.5
  Negative predictive value | 99.0
  Accuracy | 97.1

7. Secondary Outcome: Survey of the Implanting Physicians
Description: To understand the implanting physicians' experience with the implant of the Reveal LINQ, and the accompanying implanter tools. Responses to survey questions will be characterized. Below we summarize the responses to survey question "Overall, how would you rate the ease of entire implant procedure?".
Time Frame: Day of implant
Population: There have been 151 implant procedures in the study, and 151 physician implant surveys were collected. Of these 151 surveys, 149 answered the question "Overall, how would you rate the ease of entire implant procedure?".
Measure: Number; unit: Percentage of surveys
Arm/Group | Insertable Cardiac Monitor Implant
Number analyzed (Participants) | 149
Percentage of surveys
  Very Easy, No Changes Needed | 54.4
  Easy, but Needs Small Improvement | 38.9
  Needs Some Improvement | 5.4
  Needs Significant Improvement | 1.3

8. Secondary Outcome: Survey of the Patient Experience Over Time
Description: To understand the study subjects' experience with the Reveal LINQ, the patient assistant and the patient home monitor. Patient responses to survey questions will be characterized. Below we will summarize the responses to question "Based on your experience to date, please rate your satisfaction with the Reveal LINQ device" over 1 month, 6 month, and 12 month follow-up visit.
Time Frame: 12 months
Population: There were 149 patient surveys from 150 1-month follow-up visits collected, 145 surveys from 147 6-month visits, and 143 surveys from 144 12-month visits. Thus, 437 surveys were collected from 441 follow-up visits. The question "Based on your experience to date, please rate your satisfaction with the Reveal LINQ device" was answered 434 times.
Measure: Number; unit: Percentage of surveys
Units Other Than Participants: Surveys
Arm/Group | Insertable Cardiac Monitor Implant
Number analyzed (Participants) | 150
Number analyzed (Surveys) | 434
Percentage of surveys
  Very satisfied | 66.6
  Satisified | 30.2
  Needs Some Improvement | 2.8
  Needs Significant Improvement | 0.5

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Insertable Cardiac Monitor Implant
Serious Adverse Events (participants affected / at risk) | 31/151
Other Adverse Events (participants affected / at risk) | 39/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insertable Cardiac Monitor Implant (N=151)
Atrial fibrillation (Cardiac disorders) | 9 (9)
Atrial flutter (Cardiac disorders) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Implant site pain (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic tonsillitis (Infections and infestations) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Allergy test (Investigations) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insertable Cardiac Monitor Implant (N=151)
Implant Site Pain (General disorders) | 39 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less